CLINICAL TRIAL: NCT00082290
Title: Massage for the Treatment of Pain in Cancer: A Randomized Phase II Study
Brief Title: Massage Therapy in Treating Patients With Cancer Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03-046
Record Dates: First submitted 2004-05-05; First posted 2004-05-06 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2015-12

CONDITIONS: Pain; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; pain
MeSH Terms: conditions — Pain | interventions — Massage

ARMS (3):
- a massage (Experimental): About 45 minute massage
  Interventions: Other: massage therapy; Behavioral: questionaire about pain
- visit with a volunteer (Experimental): 45 minute visit
  Interventions: Other: visit with a volunteer; Behavioral: questionaire about pain
- period of quiet time (Experimental): 45 minutes of quiet time
  Interventions: Other: period of quiet time; Behavioral: questionaire about pain

INTERVENTIONS:
Other: massage therapy
  Arms: a massage
Other: visit with a volunteer
  Arms: visit with a volunteer
Other: period of quiet time
  Arms: period of quiet time
Behavioral: questionaire about pain

SUMMARY:
RATIONALE: Massage therapy may help lessen pain caused by cancer.

PURPOSE: This randomized phase II trial is studying how well massage therapy works in treating patients with cancer pain.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine whether the effects of massage therapy in patients with cancer pain are sufficiently promising to warrant a definitive trial.
* Determine the feasibility of a definitive trial.

OUTLINE: This is a randomized, controlled, pilot study. Patients are stratified according to in-patient status (yes vs no) and first baseline pain score ≥ 7 (yes vs no). Patients are randomized to 1 of 3 treatment arms.

* Arm I (massage therapy): Patients receive a light touch ("Reiki") massage over 45 minutes.
* Arm II (volunteer visit control): Patients receive a 45-minute visit from a trained volunteer who will be available to sit quietly or talk with the patient to discuss issues of concern, as desired by the patient. Volunteers will not touch the patient except to pat their shoulder or briefly hold their hand.
* Arm III (quiet time control): Patients receive 45 minutes of quiet time. Pain and mood are assessed at baseline, immediately after treatment, at 6 hours and 24 hours after treatment, and then daily for the next 5 days after treatment.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Baseline pain score ≥ 2 on a 0-10 rating scale where 0 = no pain
* Pain syndrome must be the result of cancer and/or cancer treatment

  * No postoperative or other acute procedural pain

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Concurrent pharmacologic pain therapy allowed

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2003-05; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
reduction in pain | 24 hours after treatment
  A mean change score equivalent to 2 points will be considered the minimum clinically significant reduction in pain

CONTACTS AND LOCATIONS:
Overall Officials: Barrie R. Cassileth, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States